CLINICAL TRIAL: NCT06877052
Title: Prediction of Venous Thrombosis After Fracture Operation: Comparative Analysis of Different Fracture Sites
Status: Completed | Type: Observational
Sponsor: Foshan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Qilong Nie, DIRECTOR, Foshan Hospital of Traditional Chinese Medicine
Other Study IDs: FoshanTCM User
Record Dates: First submitted 2025-03-08; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Fractures
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upper limb fracture group, lower limb fracture group, trunk fracture group, multiple fracture group

SUMMARY:
The goal of this observational study is to analyze the clinical characteristics of patients who develop lower limb deep vein thrombosis (DVT) following fracture surgery, with a focus on comparing different fracture sites. The main question it aims to answer is: How do the clinical characteristics of postoperative DVT vary across different fracture sites? The study will involve 429 patients who have been diagnosed with postoperative lower limb DVT following fracture surgery. Data will be collected on patient demographics, fracture type, surgical approach, thrombus size, number, location, and the occurrence of complications such as pulmonary embolism (PE). Participants will also be evaluated for relevant laboratory markers and clinical factors, including coagulation parameters and inflammatory markers.

By examining how these factors differ across fracture sites and their relationship to thrombus characteristics, this study seeks to better understand the risk factors and clinical course of postoperative DVT in orthopedic patients. The findings will provide valuable insights for improving patient management strategies and reducing the risk of complications such as PE in those undergoing fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age requirement: ≥18 years old, gender is not limited. (2) Including but not limited to rib fracture, femur fracture, tibia and fibula fracture, ankle fracture and other types of fracture (3) Patients with fractures who have undergone surgical treatment and patients with postoperative complications related to venous thrombosis.

  (3) The patient's clinical data (such as age, gender, fracture type, surgical method, postoperative recovery, etc.) and laboratory data (such as D-dimer, coagulation function, etc.) should be fully available.

  (4) Informed consent: Patients voluntarily participate in this study, sign informed consent, and promise to cooperate with the completion of the evaluation and follow-up in the study.

  (5) Patients with diabetes, hypertension and other comorbidities should be recorded, because these diseases may affect the occurrence of venous thrombosis.

Exclusion Criteria:

* (1) Patients with non-fracture types such as upper limb fracture and spinal fracture are not included.

  (2) Acute patients with symptoms of venous thrombosis such as deep vein thrombosis or pulmonary embolism, or patients with a history of significant thrombosis.

  (3) Patients whose clinical data or laboratory data are incomplete, resulting in no effective analysis.

  (4) Patients currently participating in other clinical trials or interventions. (5) Fracture patients who did not receive surgical treatment or only received conservative treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Demographics and Baseline Characteristics: The study population includes both male and female patients, with a focus on identifying how age, sex, and comorbid conditions may influence the development of DVT. Age ranges from 18 to over 90 years, with a significant portion of the cohort being elderly (over 60 years old), a group known to be at higher risk for thrombotic events. The patient cohort also includes individuals with varying body mass indices (BMIs), preoperative comorbidities (such as diabetes, hypertension, and cardiovascular disease), and different surgical approaches.Data Collection: For each patient, a comprehensive dataset was collected, including demographic information (age, sex, BMI), clinical characteristics (fracture type, comorbidities, type of surgical intervention), thrombus characteristics (size, location, number), and postoperative complications (e.g., the presence of pulmonary embolism). In addition, laboratory parameters, such as D-dimer levels, complete blood
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
WBC (White Blood Cell count) | From January 2024 to December 2024
  WBC (White Blood Cell count), measured in cells/µL,All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
PLT (Platelet count) | From January 2024 to December 2024
  PLT (Platelet count), measured in cells/µL; All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
ANC (Absolute Neutrophil Count) | From January 2024 to December 2024
  ANC (Absolute Neutrophil Count), measured in cells/µL; All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
Lymphocyte count | From January 2024 to December 2024
  Lymphocyte count, measured in cells/µL. All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
Activated Partial Thromboplastin Time (aPTT) | From January 2024 to December 2024
  Activated Partial Thromboplastin Time (aPTT), measured in seconds; All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
Fibrinogen | From January 2024 to December 2024
  Fibrinogen, measured in mg/dL; All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
Thrombin Time | From January 2024 to December 2024
  Thrombin Time, measured in seconds; All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
International Normalized Ratio (INR) | From January 2024 to December 2024
  International Normalized Ratio (INR), measured as a ratio,All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.

CONTACTS AND LOCATIONS:
Locations (1):
- Foshan Hospital of Traditional Chinese Medicine, Guangzhou University of Chinese Medicine, Foshan, 528051, Guangdong, China., Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Hu Y, Zhu L, Tian X, Duan F. Prevalence of preoperative deep vein thrombosis in long bone fractures of lower limbs: a systematic review and meta-analysis. J Orthop Traumatol. 2023 May 8;24(1):19. doi: 10.1186/s10195-023-00699-2. PMID 37156964
- [Background] Kobayashi T, Akiyama T, Mawatari M. Predictors of preoperative deep vein thrombosis in hip fractures: A systematic review and meta-analysis. J Orthop Sci. 2023 Jan;28(1):222-232. doi: 10.1016/j.jos.2021.08.013. Epub 2021 Sep 27. PMID 34593286